CLINICAL TRIAL: NCT06748001
Title: An Open-label, Multicenter, Rollover Study in Patients Who Participated in an Avapritinib Clinical Study
Brief Title: Avapritinib Rollover Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLU-285-2404
Record Dates: First submitted 2024-12-19; First posted 2024-12-24 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Mastocytosis, Systemic
Keywords: Indolent Systemic Mastocytosis; ISM; Advanced Systemic Mastocytosis; AdvSM; Rollover study
MeSH Terms: conditions — Mastocytosis, Systemic | interventions — avapritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Avapritinib (Experimental): Participants who have participated in a Blueprint Medicines sponsored study (the parent study) and continue to benefit from avapritinib.
  Interventions: Drug: Avapritinib

INTERVENTIONS:
Drug: Avapritinib — Avapritinib will be administered in accordance with the parent study protocol.
  Other Names: BLU-285; AYVAKIT®

SUMMARY:
The primary objective of the rollover study is to evaluate the long-term safety of avapritinib in participants who have completed a Blueprint Medicines sponsored study (parent study) and continued to benefit from avapritinib.

ELIGIBILITY:
Inclusion Criteria:

* Participated in a Blueprint Medicines sponsored avapritinib clinical study. The Sponsor reserves the right to not roll over patients who have been on drug hold for an extended time period.
* Completed End of Trial / End of Study (EOT/EOS) visit in the parent study and demonstrated compliance with the parent study requirements.
* Continue to clinically benefit from treatment with avapritinib.
* Able to give written informed consent.
* Agree to continue to use highly effective contraception as defined in this protocol.
* Female patients of childbearing potential must have negative highly sensitive serum pregnancy test within 20 days before the first dose of avapritinib. Women of nonchildbearing potential do not require this test.

Exclusion Criteria:

* Participant is participating in another interventional study.
* Participant is unwilling or unable to comply with study procedures and study restrictions.
* Participant is breastfeeding.

Other protocol-defined criteria apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events (SAEs), Adverse Events of Special Interest (AESIs), and AEs leading to Discontinuation | Up to approximately 4 years

CONTACTS AND LOCATIONS:
Locations (7):
- Universitair Ziekenhuis Antwerpen (UZA), Edegem, Belgium
- The Hospital for Sick Children, Toronto, Ontario, Canada
- A.O.U. San Giovanni di Dio e Ruggi d'Aragona di Salerno, Salerno, Italy
- Netherlands (2):
  - Universitair Medisch Centrum Groningen, Groningen
  - Erasmus Medisch Centrum, Rotterdam
- Oslo University Hospital, Oslo, Norway
- Guys and St Thomas NHS Foundation Trust - St Thomas Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No